CLINICAL TRIAL: NCT06396663
Title: The Role of the Clinical Pharmacist in Reducing Opioid Dependence at the Interface Between Hospital and Primary Care
Brief Title: DE-eSCALation of Opioids Post-surgical dischargE
Acronym: DESCALE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kent (Other)
Collaborators: Kent Community Health NHS Foundation Trust (Unknown); NHS Kent and Medway (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: University of Kent
Record Dates: First submitted 2024-04-03; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Opioid Dependence
Keywords: Prescribing; Surgery; Pain; De-escalation
MeSH Terms: conditions — Opioid-Related Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opioid de-escalation (Experimental): An early opioid deprescribing intervention, delivered by clinical pharmacists, targeting surgical patients discharged from one-of-three East Kent University Foundation Trust hospitals, with opioids.
  Interventions: Other: Rapid Opioid de-escalation; Other: Gradual Opioid de-escalation; Other: Continuation of opioids

INTERVENTIONS:
Other: Rapid Opioid de-escalation — Option 1: 10% - 50% decrease/day until opioids discontinued (≤ 10 days). For Fentanyl patches in decrements of 12 mcg/hr.
  Option 2: Stop all opioid medication completely
Other: Gradual Opioid de-escalation — Option 1: 20% - 50% decrease/weekly until opioids discontinued Option 2: 10% - 20% decrease/weekly until 30 mg daily. Then reduce by 5% - 10% everyday.
Other: Continuation of opioids — Continue on opioids and review in 1 weeks time.

SUMMARY:
The Descale Study aims to:

1. Look at the prescribing trends of opioids and the scale of long-term use following surgery within East Kent (United Kingdom)
2. Carry out a feasibility study to:

   * see if clinical pharmacists can support patients following surgery to manage their post-surgical pain safely and prevent long-term opioid use
   * calculate how much it costs the National Health Service (NHS)
   * see how the patients experienced the intervention

For Aim 1, historic records of patients who have had surgery and were discharged on opioids will be reviewed. Data collected will include type and strength of pain-relieving medication prescribed; type of surgery; number of additional opioid prescriptions following discharge; use of medical services (e.g., General Practice appointments, physiotherapy); and patient demographics.

For Aim 2, clinical pharmacists will carry out early high-risk medication safety reviews to ensure that patients have their pain managed safely. Investigators will collect key data from patients receiving the clinical pharmacist intervention to see how it affected opioid use, costs and healthcare use. Patients who took part in the study will be invited to participate in an interview and will be asked what they know about opioids and the health risks, and their experiences of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or above.
* Undergone surgery and discharged with opioid medication* less than 120mg MME/day from a participating hospital and taking it for the treatment of acute non-malignant post-surgical pain.

  * Investigators have used the British National Formulary (BNF) definition of opioids and will recruit participants who have been prescribed one or more of the following drugs: Codeine, Dihydrocodeine, Buprenorphine transdermal patches, Fentanyl transdermal patches, Morphine, Oxycodone, Tramadol, Diamorphine, Dipipanone, Tapentadol, Pentazocine.

Exclusion Criteria:

* Aged under 18 years of age.
* Unable to provide written informed consent.
* More than 90 days opioid use pre-surgery.
* On > 120 mg MME/day.
* Additional surgical procedures planned during the 3-month intervention.
* A history of methadone treatment.
* Regularly inject opioids.
* Using opioids for malignant pain.
* Undergone a caesarean section.
* Is pregnant*.
* Classified as vulnerable (e.g., severe dementia, severe co-existing or terminal medical condition).

  * Risk of miscarriage or stillbirth from opioid withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Determination of the fidelity of an early opioid deprescribing intervention led by trained clinical pharmacists in primary care and their role in the wider medicine's optimisation programme. | Month 3
  Measure the capabilities of trained clinical pharmacists to deliver an early opioid medication review by completed intervention delivery training.
Determination of the fidelity of an early opioid deprescribing intervention led by trained clinical pharmacists in primary care and their role in the wider medicine's optimisation programme. | Month 3
  Measure the capabilities of trained clinical pharmacists to deliver an early opioid medication review by observational competency checks by clinical lead.
Determination of the fidelity of an early opioid deprescribing intervention led by trained clinical pharmacists in primary care and their role in the wider medicine's optimisation programme. | Month 3
  Measure the capabilities of trained clinical pharmacists to deliver an early opioid medication review by completed medication review case reports.
Determination of the fidelity of an early opioid deprescribing intervention led by trained clinical pharmacists in primary care and their role in the wider medicine's optimisation programme. | Month 3
  Measure the capabilities of trained clinical pharmacists to deliver an early opioid medication review by the number of participants successfully deescalated.
Determination of the barriers/enablers that affect the delivery of the intervention from the perspective of the NHS stakeholders. | Up to 3 months after final follow up
  Maintain detailed records of any barriers or enablers that may occur in response to setting up the intervention and whilst delivering the intervention. Captured via Stakeholder Interviews.
Determination of the barriers/enablers that affect the delivery of the intervention from the perspective of the surgical patient. | Up to 3 months after final follow up
  Ascertain participant satisfaction of the intervention by measuring the number of participants that enrol in the study.
Determination of the barriers/enablers that affect the delivery of the intervention from the perspective of the surgical patient. | Up to 3 months after final follow up
  Ascertain participant satisfaction of the intervention by measuring the number of withdrawals from the study.
Determination of the barriers/enablers that affect the delivery of the intervention from the perspective of the surgical patient. | Up to 3 months after final follow up
  Ascertain participant satisfaction of the intervention by measuring the adherence to pharmacist medication recommendations.
Determination of the barriers/enablers that affect the delivery of the intervention from the perspective of the surgical patient. | Up to 3 months after final follow up
  Ascertain participant satisfaction of the intervention by measuring the responses to participant satisfaction questionnaire.
Determination of the barriers/enablers that affect the delivery of the intervention from the perspective of the surgical patient. | Up to 3 months after final follow up
  Ascertain participant satisfaction of the intervention by measuring the responses to participant interviews.
Establishment of the cost of delivering the intervention from the health/social care provider (NHS), perspective. | Up to 3 months after the end of recruitment
  Apply a micro-costing approach to estimate the intervention costs (combining opioid medication costs and staff costs, with Health resource use (primary care services, community-based services, hospital inpatient and outpatient services) to establish overall cost).

SECONDARY OUTCOMES:
Determination of the percentage of participants that reduce or stop opioids in 90 days | Month 3
  Measurement of the mean difference in morphine milligram equivalent (MME) dose at baseline and at 90 days.
Obtaining an understanding of trends in surgical opioid prescribing, surgical related pain, and risk factors that contribute to long term opioid use. | After the final follow up, up to 3 months
  Collect medication use data at baseline and at all follow-up appointments.
Obtaining an understanding of trends in surgical opioid prescribing, surgical related pain, and risk factors that contribute to long term opioid use. | After the final follow up, up to 3 months
  Compare opioid prescribing (type, dose, amount) at baseline for each surgical speciality and hospital.
Obtaining an understanding of trends in surgical opioid prescribing, surgical related pain, and risk factors that contribute to long term opioid use. | After the final follow up, up to 3 months
  Measure pain scores at baseline and final visits.
Obtaining an understanding of trends in surgical opioid prescribing, surgical related pain, and risk factors that contribute to long term opioid use. | After the final follow up, up to 3 months
  Measurement of risk factors in the participant population that have been previously linked to long-term opioid use, from Baseline demographics and Medical, prescription and surgical histories.
Obtaining an understanding of trends in surgical opioid prescribing, surgical related pain, and risk factors that contribute to long term opioid use. | After the final follow up, up to 3 months
  Response to Quality-Of-Life questionnaire (The EuroQol-5 Dimension (EQ5D-5L)) complete at baseline and final appointment.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Measurements of time spent finding and recruiting participants.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Measurement of number of possible surgical participants per week that could receive intervention.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Measurement of number of pharmacists available to deliver the intervention.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Measurement of number of surgical participants that accept an early Medicines Utilisation Review versus the number that are asked.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Measurement of time taken from hospital discharge to receiving first Medicines Utilisation Review.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Average time taken for each appointment.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Average time taken to successfully deescalate opioids in surgical patients.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Number of participants that are successfully deprescribed opioids within 3 months.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Number of patients that require additional appointments with the pharmacist.
Determination of the integrity, robustness, and transferability of the protocol for future adoption by the NHS. | Up to 3 months after final follow up
  Number of participants that require additional support post-90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Emma Veale, Principal Investigator — University of Kent; Dr Johanna Theron, Principal Investigator — Kent Community Health NHS Foundation Trust
Locations (1):
- Newton Place Surgery, Faversham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Jani M, Birlie Yimer B, Sheppard T, Lunt M, Dixon WG. Time trends and prescribing patterns of opioid drugs in UK primary care patients with non-cancer pain: A retrospective cohort study. PLoS Med. 2020 Oct 15;17(10):e1003270. doi: 10.1371/journal.pmed.1003270. eCollection 2020 Oct. PMID 33057368
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- See also: Public Health England, 2019. Prescribed medicines review: clinical commission group data. — http://www.gov.uk/government/publications/prescribed-medicines-review-report
- See also: Public Health England, 2019, Dependence and withdrawal associated with some prescribed medicines. — http://assets.publishing.service.gov.uk/media/5fc658398fa8f5474c800149/PHE_PMR_report_Dec2020.pdf
- See also: Office of National Statistics, 2020. Deaths related to drug poisoning in England and Wales: 2020 registrations. — http://www.ons.gov.uk/peoplepopulationandcommunity/birthsdeathsandmarriages/deaths/bulletins/deathsrelatedtodrugpoisoninginenglandandwales/2021registrations
- See also: Surgery and the NHS in numbers — http://www.rcseng.ac.uk/news-and-events/media-centre/media-background-briefings-and-statistics/surgery-and-the-nhs-in-numbers/